CLINICAL TRIAL: NCT04075084
Title: BIO|STREAM.ICM: Observation of Clinical Routine Care for Patients With BIOTRONIK Implantable Cardiac Monitors (ICMs)
Brief Title: Observation of Clinical Routine Care for Patients With BIOTRONIK Implantable Cardiac Monitors (ICMs)
Acronym: BIOSTREAM-ICM
Status: Recruiting | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: HS061
Record Dates: First submitted 2019-08-08; First posted 2019-08-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Tachycardia; Atrial Fibrillation; Syncope; Bradycardia; Cryptogenic Stroke
Keywords: Implantable Cardiac Monitor; BIOMONITOR III; BIOMONITOR IV
MeSH Terms: conditions — Tachycardia; Atrial Fibrillation; Syncope; Bradycardia; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry is performed for the long-term assessment of outcome, performance and residual safety aspects of the BIOMONITOR III and possible successors in a real-life clinical set-up. In addition, this registry is set up in a way that it may also be used as a platform for submodules to investigate additional scientific and regulatory aspects while minimizing the additional effort for the investigational sites and patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is intended to receive a BIOTRONIK Implantable Cardiac Monitor (ICM)
* Patient is able to understand the nature of the registry and to provide written informed consent.
* Patient is willing and able to use the CardioMessenger and accepts the BIOTRONIK Home Monitoring concept.

Exclusion Criteria:

* Patient is pregnant or breast feeding.
* Patient is less than 18 years old.
* Patient is participating in another interventional clinical investigation other than the submodules of BIO|STREAM.ICM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended patient population consists of all patients who would benefit from long-term cardiac rhythm monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis | The time to a relevant diagnosis can vary significantly. The time period starts with the insertion of the device.
  Device is intended to detect rare arrhythmias. Time to detect this relevant arrhythmia will be recorded.

SECONDARY OUTCOMES:
Insertion procedure and success | Data on BIOMONITOR insertion procedure and success rate are collected at day of insertion.
  Information on the insertion procedure (Operation time, handling of the BIOMONITOR incl. incision and insertion tool); Success rate of insertions.

OTHER OUTCOMES:
Sensing and noise | Data will be collected throughout the entire registry, i.e. until February 2023 (Last patient out).
  Quality of sensing Amplitude (Millivolt) and electrical noise (%) detected by the BIOMONITOR.
Inspection results of the insertion site | Data will be collected throughout the entire registry, i.e. until February 2023 (Last patient out).
  Rating of wound healing and cosmetic outcome by the physician/patient (5-level scale).
Patient contentment regarding BIOMONITOR wearability | Data will be collected throughout the entire registry, i.e. until February 2023 (Last patient out).
  Patients opinion about the wearing comfort (5-level-scale).
Device migration | Data will be collected throughout the entire registry, i.e. until February 2023 (Last patient out).
  Assessement whether the BIOMONITOR migrates under the skin.
Diagnosis and clinical actions after arrhythmia detection | Data will be collected throughout the entire registry, i.e. until February 2023 (Last patient out).
  Documentation whether the BIOMONITOR helps to detect arrhythmias. Documentation of therapies used to treat these arrhythmias and whether the BIOMONITOR helps to monitor therapy success.
Explantation / deactivation / exchange information of the BIOMONITOR | Data will be collected throughout the entire registry, i.e. until February 2023 (Last patient out).
  Collect information about explantation, deactivation and exchanges of the BIOMONITOR, such as number, reason, and data on procedure.
Adverse Events | Data will be collected throughout the entire registry, i.e. until February 2023 (Last patient out).
  Collect and analyze adverse events.
Device Deficiencies | Data will be collected throughout the entire registry, i.e. until February 2023 (Last patient out).
  Collect and analyze device deficiencies. Calculate rate (frequency) of device deficiencies.
Documentation of imaging techniques, if applied. | Data will be collected throughout the entire registry, i.e. until February 2023 (Last patient out).
  Documentation if patients underwent any MRI examinations or mammography. Documentation of exact kind of examination and occurrences with regard to the BIOMONITOR.

CONTACTS AND LOCATIONS:
Locations (31):
- Australia (2):
  - Integral Health, Adelaide
  - Royal Adelaide Hospital, Adelaide
- Nemocnice Ceske Budejovice, a.s., České Budějovice, Czechia
- France (7):
  - Hôpital Saint-André, Bordeaux
  - Le Centre Hospitalier Universitaire de Brest (CHRU Brest), Brest
  - Le Centre Hospitalier Universitaire de Caen (CHRU Caen), Caen
  - Le Centre Hospitalier Universitaire de Tours (CHRU Tours), Chambray-lès-Tours
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Haut Lévêque (CHU), Pessac
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (10):
  - St. Marienkrankhaus Klinikum Westmünsterland GmbH, Ahaus
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Rhön-Klinikum, Bad Neustadt an der Saale
  - Universitätsklinik an der Technischen Universität Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Klinikum Herford, Herford
  - Helios Health Institute GmbH, Leipzig
  - Deutsches Herzzentrum der Charité, Mitte
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Deutsches Herzzentrum der Charité, Steglitz
- Italy (2):
  - Ospedale Civile Ferrari, Castrovillari
  - Ospedale Maria Vittoria, Torino
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Portugal (2):
  - Unidade Local de Saúde do Alto Ave, E. P. E., Guimarães
  - Unidade Local de Saúde de Santa Maria, E. P. E., Lisbon
- Spain (4):
  - Centro Médico Teknon, Erandio
  - Hospital de Fuenlabrada, Fuenlabrada
  - Hospital Álvaro Cunqueiro, Vigo
  - Hospital Universitario de Araba, Vitoria-Gasteiz
- Switzerland (2):
  - GZO Spital Wetzikon, Wetzikon
  - Universitätsspital Zürich (USZ), Zurich

REFERENCES:
- [Derived] Bisignani G, De Bonis S, Pierre B, Lau DH, Hofer D, Sanfins VM, Hain A, Cabanas P, Martens E, Berruezo A, Eschalier R, Milliez P, Lusebrink U, Mansourati J, Papaioannou G, Giacopelli D, Gargaro A, Ploux S. Insertable cardiac monitor with a long sensing vector: Impact of obesity on sensing quality and safety. Front Cardiovasc Med. 2023 Mar 21;10:1148052. doi: 10.3389/fcvm.2023.1148052. eCollection 2023. PMID 37025684